CLINICAL TRIAL: NCT01809665
Title: Master Study for the MRI Compatibility of the Solia S and Solia T Pacing Lead, the Linoxsmart ProMRI and Linoxsmart ProMRI DF4 ICD (Implantable Cardioverter-defibrillator) Lead and the Corox ProMRI OTW Coronary Sinus Lead in Combination With the Ilesto/Iforia ICD or the Evia/Entovis Triple Chamber Pacemaker
Brief Title: ProMRI PROVEN Master Study
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 61
Record Dates: First submitted 2013-03-12; First posted 2013-03-13 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Safety of MR (Magnetic Resonance) Conditional CRT-pacemakers and ICDs
Keywords: ICD therapy; CRT-P therapy; MRI

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICD/CRT-P therapy: Standard indication for ICD or triple-chamber pacemaker therapy
  Interventions: Device: ICD/CRT-P therapy; Other: MRI

INTERVENTIONS:
Device: ICD/CRT-P therapy
  Other Names: Ilesto 7/5; Iforia 7/5; Evia HF-T; Entovis HF-T; Solia S; Solia T; Linoxsmart ProMRI S, SD or S DX; Linoxsmart ProMRI DF4 SD; Corox ProMRI OTW BP, -S BP or -L BP; Protego ProMRI SD
Other: MRI

SUMMARY:
This investigation is designed to provide supporting evidence for the clinical safety of the Ilesto/Iforia ICD (implantable cardioverter-defibrillator)system and the Evia/Entovis HF-T (Heart Failure) triple chamber pacemaker system when used under specific MRI (magnetic resonance imaging) conditions.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Able and willing to complete MRI testing
* Able and willing to activate and use the Cardio Messenger
* Able and willing to complete all testing required by the clinical protocol
* Available for all follow-up visits at the investigational site
* Standard indication for single, dual, or triple chamber ICD or CRT-P.
* ICD or CRT-P system to be implanted in the pectoral region
* Patient body height ≥ 140 cm
* Age ≥ 18 years

Exclusion Criteria:

* Standard contraindication for single, dual, or triple chamber ICD or CRT-P.
* Systems with an atrial lead: The patient has persistent (lasting longer than 7 days or requiring cardioversion) or permanent atrial arrhythmia
* Patient has other medical implants that may interact with MRI, e.g. abandoned pacemaker/ICD leads, lead extensions, mechanical valves, other active medical devices, non-MRI compatible devices
* Patient has other metallic artifacts / components in body that may interact with MRI
* Life expectancy of less than eight months
* Cardiac surgery in the next eight months
* Pregnant or breastfeeding
* Enrolled in another non-observational cardiac clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected for participation should be from the investigator's general patient population according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The Serious Adverse Device Effect (SADE) -free rate of the ICD/CRT-P system related to MRI | pre-MRI: approx. 2 to 5 months after implantation; post-MRI: 1 month (-2/+4 weeks) after MRI
Increase in atrial and ventricular pacing threshold(s) between pre-MRI and 1-month post-MRI | pre-MRI: approx. 2 to 5 months after implantation; post-MRI: 1 month (-2/+4 weeks) after MRI
Decrease in P-wave and R-wave amplitude (right and left) between pre-MRI and 1-month post-MRI. | pre-MRI: approx. 2 to 5 months after implantation; post-MRI: 1 month (-2/+4 weeks) after MRI

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang R. Bauer, Prof.Dr.Dr., Principal Investigator — Universitätsklinikum Würzburg, Medizinische Klinik und Poliklinik I, Oberdürrbacher Str. 6, 97080 Würzburg, Germany
Locations (23):
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Flinders Medical Center, Bedford Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Royal Adelaide Hospital, Adelaide
  - Royal Perth Hospital, Perth
  - Royal North Shore Hospital, Sydney
- Austria (2):
  - AKH Linz, Linz
  - Landesklinikum St. Pölten, Sankt Pölten
- Canada (5):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - CHUS - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Royal Alexandra Hospital, Edmonton
- University Hospital Olomouc, Olomouc, Czechia
- France (2):
  - CHU Brest, Brest
  - CHRU de Tours - Hopital Trousseau, Tours
- Germany (5):
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Coburg, Coburg
  - Elisabeth Krankenhaus Essen, Essen
  - Schwarzwald Baar Klinikum Villingen Schwenningen, Villingen-Schwenningen
  - Medizinische Universitätsklinik Würzburg, Würzburg
- Semmelweis University, Budapest, Hungary
- Stadtspital Triemli, Zurich, Switzerland